CLINICAL TRIAL: NCT04586335
Title: Open Label, Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Activity of CYH33, an Oral PI3K Inhibitor in Combination With Olaparib, an Oral PARP Inhibitor in Patients With Advanced Solid Tumors.
Brief Title: Study of CYH33 in Combination With Olaparib an Oral PARP Inhibitor in Patients With Advanced Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYH33-G102
Record Dates: First submitted 2020-08-25; First posted 2020-10-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer; Breast Cancer; Solid Tumor; Prostate Cancer; Endometrial Cancer
Keywords: PIK3CA; Olaparib
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — CYH33; olaparib

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter study which is composed of 2 parts: 1.) dose escalation and 2.) dose expansion. Bayesian optimal interval (BOIN) design will be used to determine the MTD and/or RP2D. Safety, tolerability, PK, PD, and clinical activity will also be evaluated. The CYH33 starting dose of this trial is 20 mg QD in combination with olaparib 300 mg BID. Two additional dose levels of CYH33 at 30 mg QD and 40 mg QD in combination with olaparib 200 mg BID will be evaluated. In the initial dose cohort of 20 mg CYH33 as well as in subsequent dose cohorts 20 and 30 mg QD and 40 mg QD in combination with olaparib 200 mg BID, 3 patients will be initially enrolled at each dose level of CYH33. These evaluable patients will be included into this dose level for decision making on dose selection for the next cohort. 10 mg QD of CYH33 will be evaluated in the combination with olaparib 200 mg BID, according to the BOIN design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CYH33 in Combination with Olaparib (Experimental): CYH33 in Combination with Olaparib; 20 mg CYH33 QD in combination with olaparib 300 mg BID. Additional dose levels of CYH33 at20 and 30 mg QD and CYH33 at 40 mg QD in combination with olaparib 200 mg BID will be evaluated.
  Interventions: Drug: CYH33

INTERVENTIONS:
Drug: CYH33 — Clinical Activity of CYH33, an Oral α-specific PI3K Inhibitor in Combination with Olaparib, an Oral PARP Inhibitor
  Other Names: Olaparib

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary efficacy of CYH33 in combination with olaprib in patients with DDR gene mutations and/or PIK3CA mutations, in patients who have progressed on prior PARP inhibitor, and in patients with recurrent high grade serous ovarian, fallopian tube, or primary peritoneal cancer who are platinum resistant or refractory. The study will assess if this combination will optimize anti-tumor activity, block tumor growth and overcome the resistance to PARP inhibitor treatment. The study consists 2 parts. In Part 1 dose escalation, the objective is to determine the maximum toleration dose (MTD) of the combination. The final recommended phase 2 dose (RP2D) of CYH33 in combination with olaparib will be based on the totality of an overall assessment of available safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy which could be the MTD or a dose level lower in specific cohorts of patients. In Part 2 dose expansion, the main objective is to evaluate the efficacy at RP2D.

DETAILED DESCRIPTION:
DNA damage repair (DDR) pathways can modulate cancer risk, progression and therapeutic responses. Germline mutations in genes encoding key players in the DNA-damage response (DDR), including BRCA1, BRCA2,BLM, FANCA, TP53, RAD51C, and MSH2, result in cancer susceptibility syndromes, in part because failure to adequately protect the genome against endogenous and exogenous sources of DNA damage results in the accumulation of oncogenic mutations. The mechanistic rationale for the combination of PI3K and PARP inhibitors is that PI3K inhibition leads to a downregulation of BRCA1/2 proteins, which increase the degree of HRR deficiency CYH33 is a novel, highly potent and selective inhibitor of phosphatidylinositol 3-kinase αsignificantly inhibited the activities of wild-type and mutant PI3Kα kinase as well as the specific mutant of E542K, 1047R or E545K, On July13, 2018, a Phase I first-in-human dose escalation and expansion single-agent study of CYH33 (CYH33-101) started in China (ClinicalTrials.gov identifier: NCT03544905) identify the MTD of CYH33 single agent was 40 mg. The most common treatment related adverse events (>5%) of Grade 3 was hyperglycemia. No treatment-related Grade 4 adverse event or death was reported in the ongoing trial by the cut-off date. In this combination study will assess if this combination will optimize anti-tumor activity, block tumor growth and overcome the resistance to PARP inhibitor treatment. The study consists 2 parts. In Part 1 dose escalation, the objective is to determine the maximum toleration dose (MTD) of the combination. The final recommended phase 2 dose (RP2D) of CYH33 in combination with olaparib will be based on the totality of an overall assessment of available safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy which could be the MTD or a dose level lower in specific cohorts of patients. In Part 2 dose expansion, the main objective is to evaluate the efficacy at RP2D.

ELIGIBILITY:
Key Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

1. Provide informed consent voluntarily.
2. Male and female patients ≥ 18 years of age (or having reached the age of majority according to local laws and regulations, if the age is > 18 years).
3. Patients with advanced solid tumor who have failed at least one line of prior systemic therapy or for whom standard therapy do not exist and meet the following eligibility for the corresponding part of the study:

   1. Patient must have a histologically or cytologically confirmed diagnosis of advanced recurrent or metastatic solid tumor.
   2. At least one measurable lesion as per RECIST 1.1. (Ovarian cancer participants must have measurable disease by RECIST 1.1 criteria or evaluable cancer via CA125 GCIG criteria; Prostate cancer participants must have measurable disease by RECIST 1.1 criteria or evaluable cancer via PSA response).
   3. Population eligibility:

      * Patients eligible for Part 1 dose escalation: Advanced solid tumors with any DDR gene 1) or PIK3CA 2) mutation who have failed or cannot tolerate standard treatment or currently have no standard treatment.
      * Patients eligible for Part 2 dose expansion:

        * Cohort 1: Advanced solid tumors with any selected DDR3) gene mutation
        * Cohort 2: Advanced solid tumors with PIK3CA hotspot mutation
        * Cohort 3: Advanced high grade serous ovarian, fallopian tube or primary peritoneal cancer patients with acquired PARP inhibitor resistance4)
        * Cohort 4: Advanced solid tumors with any selected DDR3) gene mutation with acquired PARP inhibitor resistance4).
        * Cohort 5: Platinum resistant/refractory5) recurrent high grade serous ovarian, fallopian tube, or primary peritoneal cancer.
4. Availability of tumor tissue sample (either fresh tumor biopsy or archival tumor tissue sample) or blood samples.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.

Key Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Patient has received any anticancer therapy (including chemotherapy, targeted therapy, hormonal therapy, biotherapy, immunotherapy, or other investigational agents.) within 28 days or 5 times of half-lives (whichever is shorter) prior to the first dose of the study treatment or who have not recovered from the side effect of such therapy.
2. Patients with contraindication to olaparib treatment or who did not tolerate olaparib previously.
3. Patients who had prior treatment with PARP inhibitor, PI3Kα inhibitor, AKT inhibitor or mTOR inhibitor (Part 2 dose expansion cohort 1& 2 only).
4. Radical radiation therapy (including radiation therapy for over 25% bone marrow) within 4 weeks prior to the first dose of the investigational product or received local palliative radiation therapy for bone metastases within 2 weeks.
5. Any toxicities from prior treatment that have not recovered to baseline or ≤ CTCAE Grade 1 before the start of study treatment, with exception of hair loss.
6. Patients with an established diagnosis of diabetes mellitus including steroid-induced diabetes mellitus.
7. Major surgery or had significant traumatic injury within 28 days prior to the first dose of the investigational product or has not recovered from major side effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 12 months
  Incidence rate of dose limiting toxicities (DLT) in the first cycle (of 28 days) of each investigated dose levels.
Tumor objective response rate (ORR) | 38 months
  Tumor objective response rate (ORR) defined as the sum of complete response (CR) and partial response (PR) as best reported by RECIST version 1.1.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 38 months
  Number, type, incidence, duration, severity and seriousness of adverse events (AEs) as assessed by CTCAE v5.0
Disease control rate (DCR) | 38 months
  Disease control rate (DCR) defined as the sum of CR, PR and stable disease (SD) by RECIST version 1.1. - Progression Free Survival (PFS).
Pharmacokinetic measures - Plasma concentration time Area Under the Curve | 12 months
  Measure the variation of CHY33/olaparib concentration in blood plasma as a function of time
Pharmacokinetic measures - Cmax | 12 months
  Measure the maximum (peak) plasma concentration(s) of CHY33/olaparib
Pharmacokinetic measures - Tmax | 12 months
  Measure of time to reach maximum (peak) plasma concentration(s) following administration of CHY33/olaparib
Pharmacokinetic measures - CL/F | 12 months
  Measure apparent total clearance(s) of CHY33/olaparib from plasma after oral administration
Pharmacokinetic measures - Vz/F | 12 months
  Measure apparent volume of distribution during terminal phase after administration of CHY33/olaparib
Pharmacokinetic measures - terminal half- life (t1/2) | 12 months
  Measure elimination half-life of CHY33/olaparib, when administered in combination

CONTACTS AND LOCATIONS:
Overall Officials: Fugen Li, PhD, Study Director — Haihe Biopharma
Locations (7):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - UT Southwestern: Simmons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Scientia Cancer Centre, Sydney, New South Wales
  - Integrated Oncology Network PTY LTD, Brisbane, Queensland
  - Monash Cancer Centre, Melbourne, Victoria
- Fudan University - Pudong Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No